CLINICAL TRIAL: NCT05975554
Title: The Effect of Low-dose Interleukin-2 on the Immune Landscape of Human Atherosclerotic Plaques at Single Cell Resolution.
Acronym: ELLIPSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Tian Zhao, BHF Clinical Lecturer in Cardiovascular Medicine., Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A096090
Record Dates: First submitted 2023-06-14; First posted 2023-08-04 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: TIA; Carotid Artery Plaque; Carotid Atherosclerosis
Keywords: Interleukin-2; IL-2; TIA; Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases | interventions — Interleukin-2

STUDY DESIGN:
Masking Description: Analysis blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose interleukin-2 (Experimental): Commercially available aldesleukin with a UK marketing authorisation will be used and will be initially prepared as per SmPC.
  Interventions: Drug: Interleukin-2 [IL-2]; Procedure: Standard care - Carotid Endarterectomy
- Control (Active Comparator): Standard of care treatment
  Interventions: Procedure: Standard care - Carotid Endarterectomy

INTERVENTIONS:
Drug: Interleukin-2 [IL-2] — 5 sequential days of treatment (1.5MIU/day subcutaneously)
  Arms: Low dose interleukin-2
Procedure: Standard care - Carotid Endarterectomy — Standard care for patients with carotid stenosis undergoing carotid endarterectomy

SUMMARY:
The goal of this clinical trail is to compare the differences in carotid plaque Treg cells' gene signature for activation, proliferation, and suppressive function using scRNA-seq in patients treated with IL-2 compared to control.

DETAILED DESCRIPTION:
Up till now our Lab has looked at Tregs and immune cells in the blood. The question remains whether low dose IL-2 can have the desired effect on Tregs in atherosclerotic plaques where they could alter the pathophysiology and potentially clinical outcomes for patients.

Up until recently, the cellular composition and cell-specific expression patterns of human atherosclerotic plaques remained elusive. However, recent breakthroughs studies using scRNA-seq, CITE-seq, and single-cell ATAC-seq on human carotid plaques have offered important insight into plaque composition, cell heterogeneity, and cell-cell interactions giving new perspectives on mechanisms of disease. The next logical stage is to use this new insight and powerful biological tool to assist in drug development for patients.

Therefore, the aims of the study are:

1. To assess if low dose IL-2, given systemically to patients at our proposed dose, can alter Tregs in atherosclerotic plaques (the disease tissue) to exhibit a proliferating, activated, and immunosuppressive phenotype
2. To assess if modulating plaque Tregs can cause a shift in the plaque immune landscape to a less inflammatory phenotype
3. To study the relationship between plaque and circulating immune cells after systemic immune modulation

ELIGIBILITY:
Inclusion Criteria:

* Presence of carotid stenosis on either ultrasound or CT scan.
* Planned to undergo carotid endarterectomy.

Exclusion Criteria:

* Autoimmune disease
* Any regular immunosuppressive treatment [Inhaled or topical steroids are permissible]
* Modified Rankin Scale score of ≥4 at screening
* Known active hepatic disease or alanine aminotransferase (ALT) > 2xULN
* Severe chronic kidney disease (defined as eGFR < 30 ml/min/1.73m2)
* Allergy or intolerance to aldesleukin
* Signs or symptoms of active infection
* History of human immunodeficiency virus (HIV), hepatitis B or C
* Current malignancy requiring active treatment
* Vaccine within 4 weeks prior to screening or plans for vaccination during study period
* Women of child-bearing potential and pregnancy
* Women who are breast-feeding
* Clinically relevant medical or surgical conditions that, in the opinion of the

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-26 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in gene expression in Tregs | Time of surgery
  Comparing differential gene expression using scRNA-seq technologies, from isolated Tregs from carotid plaques from the two patient groups (IL-2 treatment and control). Differential gene expression will be assessed using standard techniques (Z-Score)

SECONDARY OUTCOMES:
Difference in gene expression in Teff cells. | Time of surgery
  Comparing differential gene expression using scRNA-seq technologies, from isolated Teffs from carotid plaques from the two patient groups (IL-2 treatment and control). Differential gene expression will be assessed using standard techniques (Z-Score)
Immune cell gene signature, in plaque and blood. | Time of surgery
  Difference in immune cell gene signature will be compared using scRNA-seq in both plaque and blood samples, and further compared between IL-2 and control groups. Comparative analysis will be completed using gene set enrichment analysis (Enrichment Score).
Difference in gene expression patterns in Treg & Teff cells. | Baseline and at time of surgery
  Comparison between Treg and Teff cells collected at baseline and day of surgery will be compared between IL-2 and control groups. Differential gene expression will be assessed using standard techniques (Z-Score)

OTHER OUTCOMES:
Other immune cell and vascular smooth muscle cell gene expression | Time of surgery
  As per primary outcome measure but in immune cells and vascular smooth muscle cells (excluding Treg & Teff cells). Differential gene expression will be assessed using standard techniques (Z-Score)
Ligand-receptor interactions. | Time of surgery
  Differential regulation of ligand-receptor interactions between control and IL-2 treated cells will be identified by comparing single-cell/single-cell ligand-receptor interaction scores for the two groups. This measure is descriptive in nature.
T-Cell receptor profile | Time of surgery
  Difference in TCR clonality in plaques between the two groups will be assessed from clonotypes based on identical V-J gene usage and identical CDR3 junctions.
Inflammatory pathway activation. | Time of surgery
  Activation of inflammatory pathways both at plaque and systemic level. Assess for enrichment of genes involved in inflammatory pathways - enrichment score.

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrookes Hospital, Cambridge, Cambridgeshire, United Kingdom